CLINICAL TRIAL: NCT07349602
Title: The Use of Posterior Approach for Surgical Treatment of Nonspecific Spondylodiscitis.
Brief Title: Evaluation of Outcomes of Surgical Treatment for Nonspecific Infectious Spondylodiscitis Via Posterior Approach in One Center.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Organization, Federal Center for Traumatology, Orthopedics and Arthroplasty (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-2
Record Dates: First submitted 2025-11-26; First posted 2026-01-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Spondylodiscitis; Spinal Infection; Spondylitis; Discitis; Osteomyelitis; Pyogenic Infections
Keywords: pyogenic; Spondylodiscitis; posterior approach; microbiological profiles
MeSH Terms: conditions — Discitis; Spondylitis; Osteomyelitis

STUDY DESIGN:
Intervention Model Description: Patients with a deep infection affecting intervertebral discs and neighboring vertebral bodies in the thoracolumbar spine area, which were categorized as B.3.1-2 and C2-C4 according to the Pola classification.
Masking Description: Patients were informed about the upcoming surgery and its outcome - healing from infection. However, due to a lack of specialized medical training, they were unable to evaluate the use of the posterior approach. Outcome assessments were conducted without mentioning the use of the operative approach.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Posterial approach (Experimental): All patients with spondilodiscitis admitted to surgical treatment in one center. During the operation, a posterior approach was used to access the source of infection. The incision of the skin, subcutaneous fat, and aponeurosis was made with the patient in the prone position, projecting through the spinous processes of the vertebrae above the infection site and one adjacent vertebra.
  Interventions: Procedure: Posterior approach to infection site

INTERVENTIONS:
Procedure: Posterior approach to infection site — For the posterior approach, an incision through the skin, subcutaneous fat, and aponeurosis was made with the patient in the prone position, projecting through the spinous processes of the vertebrae above the infection site and one adjacent vertebra. In all cases, a thorough exploration and debridement of the infection site was performed. Bone biopsies were taken from suspected infection sites in all patients for culture.

SUMMARY:
Non-specific spondylodiscitis is a bacterial infection of the spine that in some cases requires surgical treatment. The basis of surgical treatment is the removal of affected tissues. In this case, the supportive function of the affected area is lost, which also requires stable fixation. Access to the affected part of the spine can be achieved through both anterior and posterior approaches. There is no reliable data yet confirming the advantages of each approach. Our study demonstrated successful surgical treatment of infection foci using posterior approach, no neurological or other complications were occurred. Older patients shown differences in hemoglobin levels, postoperative pain scores, the number of affected vertebrae, types of bacteria and recurrent rate.

DETAILED DESCRIPTION:
This retrospective study was conducted on 38 patients with spondylodiscitis treated using a posterior approach. Clinical data were evaluated in four age groups: under 39 years, 40-49 years, and 50-59 years and over 60.

ELIGIBILITY:
Inclusion Criteria:

- a deep infection affecting intervertebral discs and adjacent vertebral bodies in thoracolumbar spine region which were classified as B.3.1-2 and C2-C4 according to the Pola classification

Exclusion Criteria:

* cervical spine region infection
* unwilling to participate in the study,
* patients with SD of a specific etiology
* patients who received only conservative treatment,
* patients with intradural infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Surgery time | From enrollment to the end of surgery at 1 year
  Surgery time in minutes
Hospital stays | From enrollment to the end of surgery at 1 year
  Hospital stays in day
Re-operation | From enrollment to the 1-year post-surgical treatment follow-up period
  Re-operation number
Health Questionnaire EuroQol 5 Dimension five levels (EQ-5D-5L) | From enrollment to the end of surgery at 1 year
  The EQ-5D-5L descriptive system uses five dimensions and five levels of severity in each dimension. TThe five dimensions include mobility, self-care, activities of daily living, pain and discomfort, and anxiety and depression. The five levels in each dimension are worded as (1) 'not /no problems', (2) 'slight problems', (3) 'moderate problems', (4) 'severe problems' and (5) 'unable to' (mobility, self-care, usual activities), 'extreme' (pain/depression), or 'extremely' (anxiety/depression).
  Their responses are coded as a number (1, 2, 3, 4 or 5) that corresponds to the respective level of severity: 1 indicates no problems, 2-4 some problems and 3 extreme problems. In this way, a person's health state profile can be defined by a 5-digit number, ranging from 11111 (having no problems in any of the dimensions) to 55555 (having extreme problems in all the dimensions).
  The assigning of a value to an EQ-5D state is based on the time trade-off (TTO) approach.
VAS-pain after surgery | On the 2nd day after surgery
  VAS-pain on the 2nd day after surgery. Visual analog scale (0-10 VAS) and it was categorized using the following terms : no pain (0), mild (1-3), moderate (4-6), severe (7-9), or worse pain.
VAS-pain after discharge | On the 2nd day after discharge
  VAS-pain on the 2nd day after discharge. Visual analog scale (0-10 VAS) and it was categorized using the following terms : no pain (0), mild (1-3), moderate (4-6), severe (7-9), or worse pain.
Blood loss during surgery | During the intervention
  Blood loss during surgery in ml
Procalcitonin | On the 2nd day after surgery
  Procalcitonin level in the blood in ng/mL
C-reactive protein | On the 2nd day after surgery
  C-reactive protein in the blood in mg/L (Less than less than 3 mg/L consider be normal)
ESR | On the 2nd day after surgery
  Erythrocyte sedimentation rate in mm/hr. Normal ESR ; <20mm/hr.
White blood cells | On the 2nd day after surgery
  White blood cells. The normal number of WBCs in the blood is 4.5 to 11.0 × 109/L.
Hemoglobin | On the 2nd day after surgery
  Hemoglobin level in grams per deciliter. Normal hemoglobin for men ranges from 13.5 to 17.5 g/dL. Normal range for women is 12.0 to 15.5 g/dL.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal Center of Traumatology, Orthopedics and Arthroplasty, Cheboksary, Chuvashskaya Respublika, Russia

IPD SHARING:
Plan to Share IPD: Yes